CLINICAL TRIAL: NCT06180590
Title: A Prospective Cohort Study: the Efficacy of Vosevi in Treating Direct Antiviral Agent Therapy Failure Patients
Brief Title: The Efficacy of Vosevi in Treating DAA-experienced Patients
Status: Recruiting | Type: Observational
Sponsor: The Third Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: LCYJ-2023-005
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2023-06

CONDITIONS: Chronic Hepatitis C; Medication Reaction
Keywords: Vosevi; Efficacy; DAAs-experienced; Sustained Viral Response
MeSH Terms: conditions — Hepatitis C, Chronic; Drug-Related Side Effects and Adverse Reactions | interventions — Sofosbuvir; velpatasvir; voxilaprevir; sofosbuvir velpatasvir voxilaprevir drug combination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vosevi Group: Patients are administrated with once-daily oral Vosevi (Sofosbuvir/Velpatasvir/Voxilaprevir: 400mg/100mg/100mg)
  Interventions: Drug: Sofosbuvir / Velpatasvir / Voxilaprevir Oral Tablet [Vosevi]
- Sofosbuvir/Velpatasvir combined with ribavirin Group: Patients are administrated with once-daily oral Sofosbuvir/Velpatasvir (400mg/100mg) combined with ribavirin（500mg）twice a day
  Interventions: Drug: Sofosbuvir / Velpatasvir / Voxilaprevir Oral Tablet [Vosevi]

INTERVENTIONS:
Drug: Sofosbuvir / Velpatasvir / Voxilaprevir Oral Tablet [Vosevi] — Evaluate the efficacy of Vosevi in DAAs-experienced patients

SUMMARY:
Hepatitis C virus (HCV) infection remains a significant health problem in our country. The World Health Organization estimated that 71 million people worldwide had chronic HCV infection in 2015. And 399,000 people died from cirrhosis or primary hepatocellular carcinoma caused by HCV infection. In 2006, the positive rate of HCV antibody in the population aged 1-59 was 0.43%. Therefore, it was estimated that there were about 5.6 million HCV infected people in the general population, and about 10 million cases of HCV infected people in high-risk groups and high incidence areas.

Universal genotype direct antiviral agent (DAA) is the preferred antiviral therapy for hepatitis C. Sofosbuvir/velpatasvir are direct antiviral agents for hepatitis C. The results of Asian clinical trials mainly in Chinese population showed that the sustained virologic response (SVR) rates of sofosbuvir/velpatasvir at 12 weeks in genotype 1a, 1b, 2, 3a, 3b and 6 were 100%, 100%, 100%, 95%, 76% and 99%, respectively. Limited data showed that the SVR rate of sofosbuvir/velpatasvir at 12 weeks was 96% in Chinese genotype 3b patients without cirrhosis and 50% in patients with cirrhosis.

After standard antiviral therapy for hepatitis C, there are still some patients who cannot obtain SVR, and these patients are defined as DAA-experienced patients. The guidelines recommend that Sofosbuvir/Velpatasvir combined with ribavirin be used as salvage therapy for patients with DAA-experienced failure. Vosevi is a new generation of antiviral therapy for hepatitis C, which contains three components, (Sofosbuvir, Velpatasvir and Voxilaprevir. It was a salvage treatment plan for DAAs-experienced patients which was recommended by the Chinese hepatitis C prevention and treatment guidelines in 2019. However, there are insufficient data on the proportion of SVR acquired in Vosevi treated DAAs-experienced patients in Asian populations and the effectivity of antiviral therapy between Vosevi and Sofosbuvir/Velpatasvir combined with ribavirin.

In the present study, the investigators enroll DAAs-experienced hepatitis C patients. The participants are randomly divided into two groups. Then the participants are treated with Vosevi or Sofosbuvir/Velpatasvir combined with ribavirin respectively. All enrolled participants are followed-up for 3 years. Objectives of the present study are as follows:

A. To clarify the sustained virologic response rate after Vosevi therapy for DAAs-experienced patients.

B. To clarify the safety and efficacy between the Vosevi therapy and the Sofosbuvir/Velpatasvir combined with ribavirin therapy.

C. To clarify the changes of biochemistry indexes in DAAs-experienced patients after Vosevi therapy.

D. To clarify the virological relapse rate at 12 weeks after Vosevi therapy. E. To clarify the rate of cirrhosis and liver cancer during the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age of 20-70 years.
* Accepted the standard direct antiviral agent before
* HCV-RNA still positive
* Patients are administrated with once-daily oral Vosevi (Sofosbuvir/Velpatasvir/Voxilaprevir: 400mg/100mg/100mg) or Sofosbuvir/Velpatasvir (400mg/100mg) combined with ribavirin（500mg）twice a day treatment for rescue therapy.
* The good compliance of patients.

Exclusion Criteria:

* Patients with antibodies against HIV, HBV, HDV, concretion or other forms of infectious disease.
* Evidence of hepatocellular carcinoma, decompensated liver disease, auto-immune hepatitis, or significant renal, cardiovascular, respiratory or neurological comorbidity.
* Concurrent treatment with glucocorticoids, cytotoxic drugs, nonsteroidal anti-inflammatory drugs, or immune modulators.
* Pregnancy.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We enroll DAAs-experienced hepatitis C patients in The Third Affiliated Hospital of Guangzhou Medical University
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
The proportion of sustained virologic response after antiviral therapy | in one week after completed the antiviral therapy
  Testing HCV-RNA in patients after antiviral therapy using Vosevi or Sofosbuvir/Velpatasvir combined with ribavirin

SECONDARY OUTCOMES:
The proportion of ALT normalization after antiviral therapy | in one week after completed the antiviral therapy
  Testing for ALT level in patients after antiviral therapy using Vosevi or Sofosbuvir/Velpatasvir combined with ribavirin
The proportion of virologic relapse after antiviral therapy | in 12 weeks after completed the antiviral therapy
  Testing HCV-RNA in patients at 12 weeks during off-treatment
The proportion of hepatitis C patients developed into cirrhosis or liver cancer during off-treatment | Liver ultrasound every half a year after completed the antiviral therapy until the study ending
  Testing in patients every half a year during off-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xingfei Pan, PhD, Study Director — The Third Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China